CLINICAL TRIAL: NCT05152108
Title: Feasibility Clinical Study of a Novel Hybrid Brain Computer Interface for Control of Sensory-motor Coupling in Post-stroke Rehabilitation
Brief Title: Hybrid Brain Computer Interface for Control of Sensory - Motor Coupling in Post - Stroke Rehabilitation
Acronym: HYBIS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Konstantinovic Ljubica, Professor, University of Belgrade
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 6066223
Record Dates: First submitted 2021-11-13; First posted 2021-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stroke patients (Experimental): Experimental group of stroke survivors for testing the feasibility of a BCI system
  Interventions: Device: BCI feasibility test

INTERVENTIONS:
Device: BCI feasibility test — Testing the feasibility of BCI device by determining the accuracy of BCI control

SUMMARY:
HYBIS project aims to develop an innovative and unique hybrid Brain-Computer Interface (BCI) system. This BCI system is envisioned as a novel tool for targeted reinforcement of sensory motor coupling, specifically dedicated for upper-limb post-stroke rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years old at the time of enrolment
* history of cerebrovascular insult verified by computerized tomography or magnetic resonance imaging;
* stoke occurred not more than 6 months prior to study enrolment;
* subject need to be medically and neurologically stable determined by medical history and documented neurological examination;
* ability to understand, communicate and cooperate with the research team;
* ability to sit for at least 45 minutes and the ability to adhere to the study rehabilitation protocol.

Exclusion Criteria:

* any neurologic condition (beyond the stroke) or physical condition that impaired function of the affected arm
* a substantial cardiopulmonary or metabolic disorder or other major medical complication;
* history of seizures;
* moderate to severe hemispatial neglect or anosognosia involving the affected arm;
* severe sensory deficit;
* inability to understand, cooperate, and adhere to the study procedures;
* severe spasticity defined as Ashworth scale score of 4 in the affected arm;
* contraindication to stimulation system placement;
* nursing a child;
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Electrotactile BCI system accuracy | within 30 minutes after experimental session
  Electrotactile BCI system accuracy is a measure of feasibility of the prototype device. Accuracy [0 -100 %] of classification of user's mental strategy (tactile attention task towards one of the two electrical stimulation hotspots), where higher values of accuracy are related to better system control.
Motor Imagery BCI system accuracy | within 30 minutes after experimental session
  Motor Imagery BCI system accuracy is a measure of feasibility of the prototype device.
  Accuracy [0 - 100 %] of classification between rest and imaginary movement in a cue-based manner, , where higher values of accuracy are related to better system control.

SECONDARY OUTCOMES:
Fugl Meyer sensory score for upper extremity | immediately after experimental session
  Fugl Meyer sensory score for upper extremity assesses the degree of sensory impairment in the upper arm. Sensation score ranges from 0 to 12 points, divided into 4 points for light touch and 12 points for position sense. Individual items pertaining to the light touch sensation of the upper arm/ forearm and palmary surface of the hand and to the position of the shoulder/ elbow/ wrist/ thumb (IP-joint) are scored on a 3-point ordinal scale and summed for a maximum possible score of 12. The higher score is considered to represent a less sensory deficit of the subject
NASA-TLX | within 30 minutes after experimental session
  NASA Task Load Index (NASA-TLX) method assesses workload on six scales for different aspects: mental demand, physical demand, temporal demand, performance, effort, and frustration on a 21-point scale. A higher rating represents higher workload.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for rehabilitation dr Miroslav Zotovic Faculty of Medicine University of Belgrade, Belgrade, Serbia